CLINICAL TRIAL: NCT05080803
Title: Diabetic Macular Edema: Relevance of Staging Progression on Therapeutic Outcome
Status: Completed | Type: Observational
Sponsor: European School of Advanced Studies in Ophthalmology (Other)
Responsible Party: Sponsor
Other Study IDs: ESASO
Record Dates: First submitted 2021-08-11; First posted 2021-10-18 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; ESASO Classification; Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early DME: Functional results after the loading therapeutic phase. The efficacy of different drugs (bevacizumab, ranibizumab, aflibercept, desamethazone) will be analyzed separately
  Interventions: Drug: intravitreal administration of bevacizumab/ranibizumab/aflibercept/desamethazone
- Advanced DME: Functional results after the loading therapeutic phase. The efficacy of different drugs (bevacizumab, ranibizumab, aflibercept, desamethazone) will be analyzed separately
  Interventions: Drug: intravitreal administration of bevacizumab/ranibizumab/aflibercept/desamethazone
- Severe DME: Functional results after the loading therapeutic phase. The efficacy of different drugs (bevacizumab, ranibizumab, aflibercept, desamethazone) will be analyzed separately
  Interventions: Drug: intravitreal administration of bevacizumab/ranibizumab/aflibercept/desamethazone
- Atrophic diabetic maculopathy: Functional results after the loading therapeutic phase. The efficacy of different drugs (bevacizumab, ranibizumab, aflibercept, desamethazone) will be analyzed separately
  Interventions: Drug: intravitreal administration of bevacizumab/ranibizumab/aflibercept/desamethazone

INTERVENTIONS:
Drug: intravitreal administration of bevacizumab/ranibizumab/aflibercept/desamethazone — intravitreal administration

SUMMARY:
Retrospective multi-center observational study on functional and morphological outcome of initial therapy for DME according to ESASO Morphologic Classification.

DETAILED DESCRIPTION:
The ESASO morphologic classification of diabetic macular edema defines four stages of progression of the disease: early, advanced, chronic and atrophic maculopathy.

This grading is generated by the analysis of seven biomarkers that fully describe the level of retinal damage. Aim of this classification is to be a valid method for a comprehensive description of DME in scientific studies or clinical practice.

Given the recent publication of ESASO Classification, there aren't observations on the real relevance of grading DME on therapeutic outcome.

This retrospective study wants to give a preliminary answer to this important issue.

As a corollary outcome, this study will also evaluate the concordance of grading among participants.

ELIGIBILITY:
Inclusion Criteria. Eligible eyes at the retrospective review

1. Any stage of DME treated with a loading dose of 3 anti-VEGF (any type) or 1 IV dexamethasone (STEP 1).
2. OCT scans and retinal maps (radial/raster lines) at baseline (max 1 month before injection) and at one month (max 6 weeks) after the third anti-VEGF or at 3 months (max 16 weeks) after IV steroid injection (STEP 2).
3. VA at the time of both OCT examinations.

Exclusion Criteria:

1. Past ocular surgery of any kind (except for cataract surgery) or ocular pathologies other than diabetic retinopathy.
2. Macular edema considered to be due to a cause other than diabetic macular edema.
3. OCT examination suggesting that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are the primary cause of the macular edema. In the case of ERM, an OCT scan must be sent to the Coordinating Center for approval.
4. Any ocular pathology or ocular condition other than diabetes that in the opinion of the investigator might affect macular edema.
5. History of any therapy (anti-VEGF treatment, focal/grid macular photocoagulation, intravitreous or peribulbar corticosteroids) for DME or diabetic retinopathy in the past 8 months.
6. History of YAG capsulotomy performed within two months before enrollment.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: B. Major Eligibility Criteria
  1. Age ≥ 50 years
  2. Type 1 or type 2 diabetes
  3. No history/presence of any other ocular/macular pathology
  4. No history of IV/laser treatment in the past 8 months
  5. No history of cataract or other ocular surgery in the past 6 months
Sampling Method: Non-Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Functional and morphological improvement in DME after initial therapeutic loading phase, according to ESASO stage of progression of the disease. | Four months
  Visual acuity and morphological (OCT) stage of the disease (as described in ESASO DME classification) will be evaluated at time 0 and four months after the first injection of intravitreal dexamethasone or one month after the loading phase (3 monthly injections) with anti-VEGF.

SECONDARY OUTCOMES:
Validation of ESASO DME staging classification | 3 months
  After preliminary instruction on ESASO Staging system of DME, participating centers will evaluate the stage of DME at time 0 of every eye retrospectically selected to participate to the study. This staging will be than validated by the Coordinating Center, and the total concordance of staging (K index) will be used to validate the Classification

CONTACTS AND LOCATIONS:
Locations (1):
- ESASO Scientific Projects, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panozzo G, Cicinelli MV, Augustin AJ, Battaglia Parodi M, Cunha-Vaz J, Guarnaccia G, Kodjikian L, Jampol LM, Junemann A, Lanzetta P, Lowenstein A, Midena E, Navarro R, Querques G, Ricci F, Schmidt-Erfurth U, Silva RMD, Sivaprasad S, Varano M, Virgili G, Bandello F. An optical coherence tomography-based grading of diabetic maculopathy proposed by an international expert panel: The European School for Advanced Studies in Ophthalmology classification. Eur J Ophthalmol. 2020 Jan;30(1):8-18. doi: 10.1177/1120672119880394. Epub 2019 Nov 12. PMID 31718271
- [Background] Panozzo G, Mura GD, Franzolin E, Giannarelli D, Albano V, Alessio G, Arrigo A, Casati S, Cassottana P, Contardi C, D'Aloisio R, Fasce F, Gusson E, Marchini G, Mastropasqua L, Niccolo M, Palmisano C, Pastore MR, Saviano S, Tognetto D, Bandello F. Early DMO: a predictor of poor outcomes following cataract surgery in diabetic patients. The DICAT-II study. Eye (Lond). 2022 Aug;36(8):1687-1693. doi: 10.1038/s41433-021-01718-4. Epub 2021 Aug 3. PMID 34345028